CLINICAL TRIAL: NCT06676059
Title: SMART-r: Substance Monitoring and Active Relapse Tracking Repository
Status: Recruiting | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002094; 002094-DA
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-03-27

CONDITIONS: Alcoholism; Substance-Related Disorders
Keywords: Alcohol; Substance use; digital phenotyping
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults who use substances: Adults 18 years or older who use drugs or alcohol

SUMMARY:
Background:

About 1.5 million adults in the US enter alcohol or substance use treatment programs each year. Unfortunately, more than half of patients do not finish their program. For those who start treatment, about 70% return to substance use within weeks or months after starting treatment. To discover why patients drop out of treatment and return to substance use - and what can be done about it - researchers need to learn more about people who use drugs and alcohol.

Objective:

To create a data repository by gathering survey and smartphone data from adults who use drugs and alcohol in order to conduct future research.

Eligibility:

Adults who have used drugs or alcohol in the past and have a Android smartphone. The researchers will recruit targeted demographics at different times throughout the duration of the study period.

Design:

Data will be collected for up to 6 months. All research activities will be online.

Participants will download a smartphone app called TTRU-Curtis AWARE and keep it active on their phone. The app will run in the background and collect participant data, including: screen unlocks, duration of time the screen is on; apps used; words typed (except passwords); duration and time of phone calls; estimated location (exact location is not collected); and movement, such as how many steps are taken in a day. All personally identifying information is automatically removed before the data is stored (including phone numbers, names, or locations described in messages).

Each day, participants will receive a text with a link to a survey. They will answer questions about their mood, behavior, and substance use from the day before. This survey should take less than 5 minutes to complete.

Every 30 days, participants will complete a longer survey. They will answer questions about their personal relationships, risky behaviors, mood, substance use, and feelings. They can skip any questions they do not feel comfortable answering. These surveys should take about 30 minutes to complete.

Participants may opt to allow researchers to access their social media posts.

DETAILED DESCRIPTION:
Description:

This project aims to establish a comprehensive data repository for conducting secondary research, including the analysis of digital phenotype data from individuals who have historically used drugs, including alcohol. Our hypothesis is that digital phenotyping can reveal unique behavioral patterns and risk factors associated with substance use. By collecting data such as smartphone app usage, social media interactions, phone sensor measurements, and wearable device metrics, the TTRU research lab will be able to conduct secondary analyses and uncover insights that could inform prevention and intervention strategies with individuals who use substances.

Objectives

Primary Objective:

The primary objective is to establish the NIDA-IRP Technology and Translational Research Unit (TTRU) Substance Monitoring and Active Relapse Tracking Repository (SMART-r) for collection, storage, and analysis of the human data from individuals who use substances. The secure, high-quality resource of digital, sensor, social media, self-report, and clinical data (Repository Materials) will be created. Core variables of interest include sensor data, language, and relevant self-report measures. The intention to collect digital phenotyping data is to aid in the efficiency and efficacy of secondary research investigating health outcomes for individuals who use substances by creating a repository of de-identified data.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in the repository, an individual must meet all of the following criteria:

* Must understand and be willing to complete an online informed consent process.
* Be an adult aged 18 or older.
* Self-report alcohol or other drug use within the past 30 days.
* Have an Android smartphone as their primary mobile phone.

  --The TTRU-CURTIS AWARE App does not have iPhone iOS functionality.
* Have a minimum of 500 sent text messages and 1000 words exchanged through SMS (text messages).
* Be willing to adhere to the procedures, including downloading the AWARE app onto their smartphone and keeping it active throughout the data collection period, completing baseline questionnaires, daily diary EMAs, and follow-up surveys.
* Understand and write in English.

  --This exclusion criterion is included because future research on the data collected will include linguistic analysis. all linguistic analyses, we remove rare words (e.g., words must be said by at least 95% of participants). Additionally, there are cultural differences across languages and, thus, interpreting language results across more than one language becomes difficult. As a result, we must keep analysis limited to a single language (English), since words in other languages will not meet that criteria.
* Live in the United States.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this repository:

-Any impairment severe enough to preclude informed consent or valid self-report.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have used drugs or alcohol in the past and have a Android smartphone. The researchers will recruit targeted demographics at different times throughout the duration of the study period.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2044-12-31 (Estimated); Study Completion 2044-12-31 (Estimated)

PRIMARY OUTCOMES:
SMARTr data repository | 20 years
  The primary objective is to establish the NIDA-IRP Technology and Translational Research Unit (TTRU) Substance Monitoring and Active Relapse Tracking Repository (SMART-r) for collection, storage, and analysis of the human data from individuals who use substances.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda L Curtis, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregated data will be made available upon request.

REFERENCES:
- [Background] Sinha R. New findings on biological factors predicting addiction relapse vulnerability. Curr Psychiatry Rep. 2011 Oct;13(5):398-405. doi: 10.1007/s11920-011-0224-0. PMID 21792580
- [Background] Bauer LO. Predicting relapse to alcohol and drug abuse via quantitative electroencephalography. Neuropsychopharmacology. 2001 Sep;25(3):332-40. doi: 10.1016/S0893-133X(01)00236-6. PMID 11522462
- [Background] Claus RE, Kindleberger LR. Engaging substance abusers after centralized assessment: predictors of treatment entry and dropout. J Psychoactive Drugs. 2002 Jan-Mar;34(1):25-31. doi: 10.1080/02791072.2002.10399933. PMID 12003110
- [Background] Darke S, Campbell G, Popple G. Retention, early dropout and treatment completion among therapeutic community admissions. Drug Alcohol Rev. 2012 Jan;31(1):64-71. doi: 10.1111/j.1465-3362.2011.00298.x. Epub 2011 Mar 22. PMID 21426420
- [Background] Evans E, Li L, Hser YI. Client and program factors associated with dropout from court mandated drug treatment. Eval Program Plann. 2009 Aug;32(3):204-12. doi: 10.1016/j.evalprogplan.2008.12.003. Epub 2008 Dec 11. PMID 19150133
- [Background] Lejuez CW, Zvolensky MJ, Daughters SB, Bornovalova MA, Paulson A, Tull MT, Ettinger K, Otto MW. Anxiety sensitivity: a unique predictor of dropout among inner-city heroin and crack/cocaine users in residential substance use treatment. Behav Res Ther. 2008 Jul;46(7):811-8. doi: 10.1016/j.brat.2008.03.010. Epub 2008 Mar 28. PMID 18466878
- [Background] Lopez-Goni JJ, Fernandez-Montalvo J, Arteaga A. Addiction treatment dropout: exploring patients' characteristics. Am J Addict. 2012 Jan-Feb;21(1):78-85. doi: 10.1111/j.1521-0391.2011.00188.x. Epub 2011 Dec 1. PMID 22211350
- [Background] Odenwald M, Semrau P. Dropout among patients in qualified alcohol detoxification treatment: the effect of treatment motivation is moderated by Trauma Load. Subst Abuse Treat Prev Policy. 2013 Mar 21;8:14. doi: 10.1186/1747-597X-8-14. PMID 23514277
- [Background] Epstein DH, Marrone GF, Heishman SJ, Schmittner J, Preston KL. Tobacco, cocaine, and heroin: Craving and use during daily life. Addict Behav. 2010 Apr;35(4):318-24. doi: 10.1016/j.addbeh.2009.11.003. Epub 2009 Nov 12. PMID 19939575
- [Background] Epstein DH, Willner-Reid J, Vahabzadeh M, Mezghanni M, Lin JL, Preston KL. Real-time electronic diary reports of cue exposure and mood in the hours before cocaine and heroin craving and use. Arch Gen Psychiatry. 2009 Jan;66(1):88-94. doi: 10.1001/archgenpsychiatry.2008.509. PMID 19124692
- [Background] Preston KL, Vahabzadeh M, Schmittner J, Lin JL, Gorelick DA, Epstein DH. Cocaine craving and use during daily life. Psychopharmacology (Berl). 2009 Dec;207(2):291-301. doi: 10.1007/s00213-009-1655-8. Epub 2009 Sep 24. PMID 19777216
- [Background] Koob G, Kreek MJ. Stress, dysregulation of drug reward pathways, and the transition to drug dependence. Am J Psychiatry. 2007 Aug;164(8):1149-59. doi: 10.1176/appi.ajp.2007.05030503. PMID 17671276
- [Background] McHugh RK. Treatment of co-occurring anxiety disorders and substance use disorders. Harv Rev Psychiatry. 2015 Mar-Apr;23(2):99-111. doi: 10.1097/HRP.0000000000000058. PMID 25747923
- [Background] Berenz EC, Coffey SF. Treatment of co-occurring posttraumatic stress disorder and substance use disorders. Curr Psychiatry Rep. 2012 Oct;14(5):469-77. doi: 10.1007/s11920-012-0300-0. PMID 22825992
- [Background] Crosby R, Holtgrave DR, Stall R, Peterson JL, Shouse L. Differences in HIV risk behaviors among black and white men who have sex with men. Sex Transm Dis. 2007 Oct;34(10):744-8. doi: 10.1097/OLQ.0b013e31804f81de. PMID 17565334
- [Background] Millett GA, Peterson JL, Wolitski RJ, Stall R. Greater risk for HIV infection of black men who have sex with men: a critical literature review. Am J Public Health. 2006 Jun;96(6):1007-19. doi: 10.2105/AJPH.2005.066720. Epub 2006 May 2. PMID 16670223
- [Background] Levy ME, Wilton L, Phillips G 2nd, Glick SN, Kuo I, Brewer RA, Elliott A, Watson C, Magnus M. Understanding structural barriers to accessing HIV testing and prevention services among black men who have sex with men (BMSM) in the United States. AIDS Behav. 2014 May;18(5):972-96. doi: 10.1007/s10461-014-0719-x. PMID 24531769
- [Background] Shuper PA, Joharchi N, Bogoch II, Loutfy M, Crouzat F, El-Helou P, Knox DC, Woodward K, Rehm J. Alcohol consumption, substance use, and depression in relation to HIV Pre-Exposure Prophylaxis (PrEP) nonadherence among gay, bisexual, and other men-who-have-sex-with-men. BMC Public Health. 2020 Nov 25;20(1):1782. doi: 10.1186/s12889-020-09883-z. PMID 33256651
- [Background] Gebru NM, Benvenuti MC, Rowland BHP, Kalkat M, Chauca PG, Leeman RF. Relationships among Substance Use, Sociodemographics, Pre-Exposure Prophylaxis (PrEP) Awareness and Related Attitudes among Young Adult Men Who Have Sex with Men. Subst Use Misuse. 2022;57(5):786-798. doi: 10.1080/10826084.2022.2040030. Epub 2022 Feb 21. PMID 35188880
- [Background] Crozier ME, Farokhnia M, Persky S, Leggio L, Curtis B. Relationship between self-stigma about alcohol dependence and severity of alcohol drinking and craving. BMJ Ment Health. 2023 Nov 22;26(1):e300852. doi: 10.1136/bmjment-2023-300852. PMID 37993282
- [Background] Shiffman S. Ecological momentary assessment (EMA) in studies of substance use. Psychol Assess. 2009 Dec;21(4):486-97. doi: 10.1037/a0017074. PMID 19947783
- [Background] Torous J, Onnela JP, Keshavan M. New dimensions and new tools to realize the potential of RDoC: digital phenotyping via smartphones and connected devices. Transl Psychiatry. 2017 Mar 7;7(3):e1053. doi: 10.1038/tp.2017.25. PMID 28267146
- [Background] Jain SH, Powers BW, Hawkins JB, Brownstein JS. The digital phenotype. Nat Biotechnol. 2015 May;33(5):462-3. doi: 10.1038/nbt.3223. No abstract available. PMID 25965751
- [Background] Barnett I, Torous J, Staples P, Sandoval L, Keshavan M, Onnela JP. Relapse prediction in schizophrenia through digital phenotyping: a pilot study. Neuropsychopharmacology. 2018 Jul;43(8):1660-1666. doi: 10.1038/s41386-018-0030-z. Epub 2018 Feb 22. PMID 29511333
- [Background] Boukhechba M, Chow P, Fua K, Teachman BA, Barnes LE. Predicting Social Anxiety From Global Positioning System Traces of College Students: Feasibility Study. JMIR Ment Health. 2018 Jul 4;5(3):e10101. doi: 10.2196/10101. PMID 29973337
- [Background] Giorgi S, Yaden DB, Eichstaedt JC, Ungar LH, Schwartz HA, Kwarteng A, Curtis B. Predicting U.S. county opioid poisoning mortality from multi-modal social media and psychological self-report data. Sci Rep. 2023 Jun 3;13(1):9027. doi: 10.1038/s41598-023-34468-2. PMID 37270657
- [Background] Son Y, Clouston SAP, Kotov R, Eichstaedt JC, Bromet EJ, Luft BJ, Schwartz HA. World Trade Center responders in their own words: predicting PTSD symptom trajectories with AI-based language analyses of interviews. Psychol Med. 2023 Feb;53(3):918-926. doi: 10.1017/S0033291721002294. Epub 2021 Jun 22. PMID 34154682
- [Background] Meyerhoff J, Liu T, Stamatis CA, Liu T, Wang H, Meng Y, Curtis B, Karr CJ, Sherman G, Ungar LH, Mohr DC. Analyzing text message linguistic features: Do people with depression communicate differently with their close and non-close contacts? Behav Res Ther. 2023 Jul;166:104342. doi: 10.1016/j.brat.2023.104342. Epub 2023 May 27. PMID 37269650